CLINICAL TRIAL: NCT00580918
Title: Functional MRI Study of Attention in Normal Controls and Traumatic Brain Injured Patients
Status: Withdrawn | Type: Observational
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: HS#2003-3139
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury; fMRI
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Mild Traumatic Brain Injury group
  Interventions: Other: functional magnetic resonance imaging fMRI
- 2: Normal healthy control group
  Interventions: Other: functional magnetic resonance imaging fMRI

INTERVENTIONS:
Other: functional magnetic resonance imaging fMRI — functional magnetic resonance imaging fMRI

SUMMARY:
The purpose of this study will be to assess the attentional ability of patients with mild to moderate traumatic brain injury (TBI) using the functional Magnetic Resonance Imaging (fMRI) technique. Methodology for specific aim 1: sagittal pilot scan, 3-D anatomical MRI, Whole brain echo-planar imaging (EPI), and functional MRI techniques with traumatic brain injured subjects doing a Continuous Performance Test (CPT) attention task and compare the pattern of activation with those of normal controls to see if there is a failure to activate frontal lobes in the traumatic brain injured subjects.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate brain injury patients referred to the UCI Brain Imaging Center.

  * Mild brain injury patients will be defined as having a Glascow Coma Scale (GCS) scale of 13-15.
  * Moderate brain injury brain injury patients will be defined as having a Glascow Coma Scale (GCS) scale of 9-12 .
* Normal healthy control subjects (20)

Exclusion Criteria:

* Pre-accident neuropathology, psychopathology, or secondary neuropathological complications, or chemical abuse
* Patients who required intracranial surgical intervention
* Children, pregnant women, or institutionalized individuals unable to freely give consent
* Patients with implanted surgical clips (hemostatic clips) or other ferromagnetic material
* Patients engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials, or who may have imbedded metal fragments from military activities
* Patients with permanent (tattoo) eye-liner or with facial make-up (severe eye irritation has been reported)
* Patients with metallic implants, because they may cause artifacts in diagnostic images due to magnetic field distortion
* Patients with implanted prosthetic heart valves
* Patients with pacemakers, neuro-stimulation devices
* Subjects who have severe claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mild Traumatic Brain Injury Normal health controls
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-10; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
fMRI scans | three to four years post injury

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Wu, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States